CLINICAL TRIAL: NCT02818400
Title: Composite Tissue Allotransplantation of the Face: Anatomical and Functional Evaluation
Acronym: AFTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHRCN06-PR-DEVAUCHELLE
Record Dates: First submitted 2016-06-10; First posted 2016-06-29 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Surgery, Oral
Keywords: maxillofacial surgery; face graft; composite tissue; stem cell infusion; allotransplantation; microsurgery
MeSH Terms: interventions — Vascularized Composite Allotransplantation

ARMS (1):
- Composite tissue allotransplantation (Experimental)
  Interventions: Procedure: composite tissue allotransplantation

INTERVENTIONS:
Procedure: composite tissue allotransplantation

SUMMARY:
In hindsight, the first "face graft" raises the fundamental problem of composite tissue allotransplantation (hand, larynx, abdominal wall, etc.) with the addition of specific technical and philosophical problems.

By proposing a prospective study concerning five new patients over the next three years, in the light of this first experience, the authors would like to confirm the surgical feasibility of this type of procedure, possibly extending it to other parts of the face (lateral third) and, like English and American teams, considering the possibility of total facial surface reconstruction.

In parallel, and while complying with the usual immunosuppression procedures, the deliberate choice of creating a microchimerism by the infusion of bone marrow stem cells (the origin and quantity of which will need to be determined) will be reaffirmed, in order to improve mucocutaneous tissue tolerance, while confirming the safety of this type of approach.

Five new cases will also provide observations for the many new fields of research developing around composite tissue transplants (neurophysiology, skin histopathology, psychiatry, haematology, immunology, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients with loss of unrepairable substance by conventional techniques shreds, at the front

Exclusion Criteria:

* Facial lesions repaired by conventional reconstructive surgery techniques
* History of malignancy in remission for less than 5 years
* Malignant neoplasm undergoing changes
* Severe psychiatric history
* Patients above a score of 2 on the scale of the ASA (American Society of Anesthesiology)
* Patients above a grade 1 in the classification NYHA ( New York Heart Association )
* insufficient with renal creatinine clearance less than 70 mL / min or presence of a proteinuria
* Severe hypertension

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2009-11; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
functional recovery : motor recovery | 1 year
  labial contact allowing complete mouth closure
functional recovery : sensory recovery | 1 year
  Sensitivity to light touch, as assessed with the use of static monofilaments
functional recovery : sensory recovery | 1 year
  sensitivity to heat and cold

SECONDARY OUTCOMES:
functional recovery : motor recovery | 2 years, 5 years
  labial contact allowing complete mouth closure
functional recovery : sensory recovery | 2 years, 5 years
  Sensitivity to light touch, as assessed with the use of static monofilaments
functional recovery : sensory recovery | 2 years, 5 years
  sensitivity to heat and cold

CONTACTS AND LOCATIONS:
Overall Officials: Bernard DEVAUCHELLE, Md, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France